CLINICAL TRIAL: NCT06521320
Title: Speaking Valve Combined With Airway Pressure Predicts Upper Airway Patency in Adult Tracheotomized Patients: a Prospective Cohort Study
Brief Title: Speaking Valve Combined With Airway Pressure Predicts Upper Airway Patency in Adult Tracheotomized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jingyi Ge, Principal Investigator, Capital Medical University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2021Z-001
Record Dates: First submitted 2024-07-12; First posted 2024-07-25 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-09

CONDITIONS: Tracheotomy
Keywords: upper airway patency; speaking valve; upper airway; prolonged tracheostomized patients; transtracheal end-expiratory pressure
MeSH Terms: interventions — Bronchoscopy

STUDY DESIGN:
Intervention Model Description: All patients were given a speaking valve combined with airway pressure measurement and bronchoscopy.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Upper airway patency (Experimental): Upper airway patency confirmed by speaking valve combined with airway pressure measurement or bronchoscopy
  Interventions: Diagnostic Test: speaking valve combined with airway pressure; Diagnostic Test: Bronchoscopy
- Upper airway obstruction (Experimental): Upper airway obstruction confirmed by speaking valve combined with airway pressure measurement or bronchoscopy
  Interventions: Diagnostic Test: speaking valve combined with airway pressure; Diagnostic Test: Bronchoscopy

INTERVENTIONS:
Diagnostic Test: speaking valve combined with airway pressure — All patients were given speaking valves and airway pressure was measured to assess upper airway patency.
Diagnostic Test: Bronchoscopy — The same examiner performed bronchoscopy on all patients to assess upper airway patency.

SUMMARY:
This study was aimed to evaluate whether speaking valve combined with airway pressure could predict upper airway patency non-invasively in prolonged tracheostomized patients, identify candidates who need following endoscopy examination.

DETAILED DESCRIPTION:
Tracheotomy is an effective means of treating critically ill patients, but its postoperative management faces many challenges, especially in the assessment and monitoring of upper airway patency. Although the indwelling tracheostomy tube plays an important role in maintaining airway patency and assisting breathing, it may also cause a series of complications, including airway stenosis, granulation tissue hyperplasia, airway collapse, and laryngeal dysfunction. The patency of the upper airway after tracheotomy is directly related to the patient's spontaneous breathing ability and quality of life. Although the existing bronchoscopy provides accurate diagnostic information, its invasiveness and high cost limit its application in extensive and high-frequency monitoring. Finding a non-invasive, easy-to-operate and accurate alternative method is of great clinical significance.The speaking valve is a one-way valve placed at the end of the tracheostomy tube that directs airflow to the upper airway when the cuff is deflated. Airway pressure measurement is a simple, non-invasive method that measures the pressure inside the tracheostomy tube to infer airway patency and resistance levels. Combining the two for a systematic assessment of upper airway patency in tracheostomy patients may provide a new, efficient, non-invasive monitoring tool for the clinic. By comparing the results of speaking valve combined with airway pressure measurement with the "gold standard" bronchoscopy results, its sensitivity and accuracy in assessing upper airway patency are verified, which is expected to not only provide a non-invasive, easier-to-use bedside assessment tool, but also improve the quality of patient care and their quality of life. Our hospital's respiratory rehabilitation center has the appropriate infrastructure and professional staffing to conduct research safely and in a standardized manner.

ELIGIBILITY:
Inclusion Criteria:

* Weaned from ventilator more than 48 hours
* No any organ failure
* No sepsis
* Stable heart rate and blood pressure
* Lung infection under control
* PCO2<60mmHg
* Patient and family sign informed consent form

Exclusion Criteria:

* Serious dysfunction of vital organs
* Unable tolerance of cuff deflated
* Laryngopharyngeal trauma
* Known severe upper airway obstruction before referrer to our department
* Endoscopy(bronchoscopy or laryngoscopy) has been performed and the condition of the upper airway has known

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Upper airway patency | The patients started using the speaking valve combined with airway pressure measurement on the day of enrollment. After that, bronchoscopy should be performed within 48 hours.
  Speaking valve combined with airway pressure protocol: After suction of oral and nasal secretion, the cuff was deflated. Then the speaking valve was placed. Supplement oxygen could be provided from nose. Connect a pressure measuring device for airway pressure. Then the tracheostomy tube was downsized according to patient's status (This decision was decided by a multidisciplinary team through consultation). Patients who could tolerate speaking valve and airway pressure<10cmH2O were assumed Upper airway patency group. Patients who cannot tolerate the speaking valve or whose airway pressure is ≥10cmH2O even after downsizing the tracheostomy are in the Upper airway obstruction group.
  Bronchoscopy protocol: Use bronchoscopy through nose to observe the upper airway through the glottis and around the cuff. Patients with bilateral vocal cord distance <3 mm or Cotton grade II or above were considered to have upper airway obstruction during bronchoscopy evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Jingyi Ge, Principal Investigator — specify unaffiliated
Locations (1):
- Beijing Rehabilitation Hospital of Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No